CLINICAL TRIAL: NCT03485807
Title: The Virginia Commonwealth University (VCU) Stress Reduction Study
Brief Title: Stress Reduction Training for Emotion Regulation and Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HM20012124
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Stress Reduction
Keywords: stress; mindfulness; active coping

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Training (MT) (Experimental)
  Interventions: Behavioral: Mindfulness Training (MT)
- Active Coping Training (CT) (Experimental)
  Interventions: Behavioral: Active Coping Training (CT)

INTERVENTIONS:
Behavioral: Mindfulness Training (MT) — 2 week SmartPhone-based mindfulness training
  Arms: Mindfulness Training (MT)
Behavioral: Active Coping Training (CT) — 2 week SmartPhone-based structurally equivalent coping training
  Arms: Active Coping Training (CT)

SUMMARY:
This study will examine whether stress reduction training - which a growing body of research indicates has manifold benefits for behavior regulation, emotion regulation, and other salutary outcomes of relevance to this proposal - predicts lab-based and daily life-based neural and behavioral outcomes indicative of reduced stress, including emotions, desires, and reactions to adverse events such as social conflict.

DETAILED DESCRIPTION:
This research study seeks to understand how stress reduction training influences neural responses (brain activation) and behavior related to stress, including emotions, desires, and reactions to adverse events such as social conflict. The full research project will be conducted over approximately 4-6 weeks, and will consist of two data collection sessions on the Virginia Commonwealth University (VCU) campus, one before and one after a 14-day stress reduction training course conducted via mobile phone (SmartPhone). The two courses entail instructor-facilitated stress reduction exercises previously shown to reduce stress and improve well-being. Participants will be randomly assigned to a mindfulness course or an active coping course. Both of these courses - mindfulness training (MT) and coping training (CT) - involve expert-facilitated mental wellness techniques. MT emphasizes mindfulness-based techniques to reduce stress and promote well-being, whereas CT emphasizes established emotion regulation techniques to reduce stress and promote well-being.

Some study details are purposely omitted at this time to preserve scientific integrity.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking (will not be advertised but screened)
2. Stable medication regiment for 8 weeks prior to enrollment if taking antidepressant or anxiolytic medications. (will not be advertised but screened)
3. Free of major, uncorrected sensory impairments and cognitive deficits
4. Free of a certain psychiatric disorders or history thereof; specifically, a new diagnosis of a (non-acute) medical or psychiatric condition within the last 3 months, report a hospitalization over the last 3 months, report current drug abuse (e.g., recreational drug use, alcohol intake in excess of 2 drinks per day).
5. Personal SmartPhone (Android or Apple operating systems).

Exclusion Criteria:

1. non-English speaking
2. are unwilling or unable to complete study assessments or treatments
3. present fMRI safety risks (e.g., ferromagnetic implants, body weight > 300 lbs)
4. report a new diagnosis of a (non-acute) medical or psychiatric condition within the last 3 months
5. report a hospitalization over the last 3 months
6. report current drug abuse (e.g., recreational drug use, smoke more than ½ pack per day, alcohol intake in excess of 2 drinks per day)
7. are prisoners or pregnant women
8. no personal SmartPhone (Android or Apple operating systems)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Level of lab-based emotion regulation (behavior) | Baseline, post-test (within 3 weeks after intervention)
  Measured by affective face matching task

SECONDARY OUTCOMES:
Neural activation associated with emotion regulation | Baseline, post-test (within 3 weeks after intervention)
  Measured by functional magnetic resonance imaging (fMRI) during affective face matching task
Change in level of stress, desires, social conflict in daily life | Baseline, post-test (within 3 weeks after intervention)
  Measured by ecological momentary assessments of stress, desires, social interactions

CONTACTS AND LOCATIONS:
Overall Officials: Kirk W Brown, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Rahrig H, Bjork JM, Tirado C, Chester DS, Creswell JD, Lindsay EK, Penberthy JK, Brown KW. Punishment on Pause: Preliminary Evidence That Mindfulness Training Modifies Neural Responses in a Reactive Aggression Task. Front Behav Neurosci. 2021 Jul 23;15:689373. doi: 10.3389/fnbeh.2021.689373. eCollection 2021. PMID 34366804

DOCUMENTS (1):
  • Informed Consent Form (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT03485807/ICF_000.pdf